CLINICAL TRIAL: NCT02889016
Title: Neurobiologic, Immunologic, and Rheumatologic Markers in Youth With PANS
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jennifer Frankovich, Clinical Associate Professor, Stanford University
Other Study IDs: 26922
Record Dates: First submitted 2016-08-22; First posted 2016-09-05 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Pediatric Acute-Onset Neuropsychiatric Syndrome; Pediatric Autoimmune Neuropsychiatric Disorders Associated With Streptococcal Infections; PANS; PANDAS
Keywords: PANS; PANDAS
MeSH Terms: conditions — Pediatric acute-onset neuropsychiatric syndrome; Pediatric Autoimmune Neuropsychiatric Disorders Associated with Streptococcal infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood mononuclear cells (PBMCs) are collected from patients during flares and remissions. Samples will be used for genome-wide association studies (GWAS), time-of-flight mass spectrometry (CyTOF), TCR analyses, antibody profiling, and monocyte characterizations.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PANS group: 500 children, 1-18 years old at onset with a strict diagnosis of PANS/PANDAS will be recruited
- Health Controls: 100 healthy children age- and gender- matched to the PANS group will be recruited

SUMMARY:
This study is an investigation of the neurologic, immunologic, and rheumatologic markers of Pediatric Acute-Onset Neuropsychiatric Syndrome (PANS). PANS is a condition characterized by the abrupt, dramatic onset of obsessive compulsive disorder (OCD) and/or eating restriction accompanied by equally abrupt and severe co-morbid neuropsychiatric symptoms, which include anxiety, emotional lability, depression, irritability, aggression, oppositionality, deterioration in school performance, behavioral (developmental) regression, sensory amplification, movement abnormalities, sleep disturbance, and urinary frequency. PANS is thought to be caused by infection, inflammation, or alternate triggers that is associated with a brain response that leads to these symptoms. The purpose of this study is to examine specific neurologic, immunologic, rheumatologic, and genomic, components in children with the acute-onset of psychiatric symptoms. This research may begin to uncover a much larger story of autoimmune processes that are involved in psychiatric disorders of childhood. By better understanding the etiologic components of psychiatric phenomenon, future treatments may be better targeted to underlying causes.

DETAILED DESCRIPTION:
The investigators will recruit 500 children, 1-18 years old at onset with PANS/PANDAS. They will be treatment naive and within one month of onset/exacerbation. The 500 children with PANS will be gender- and age-matched to 100 healthy children, to allow examination of immunologic, neurologic, genomic, and behavioral differences between these two groups of children.

ELIGIBILITY:
Inclusion Criteria:

* Children with PANS

  1. Age 1-18 at onset of PANS
  2. Diagnosis of PANS: abrupt onset of OCD or food restriction, and at least two of the following associated symptoms: frequent urination, worsening handwriting/cognition, inattention, anorexia, separation anxiety, oppositionality, irritability/rage outbursts, and emotional lability.
  3. Patients must live within 90 miles of Stanford University and have a new onset of PANS illness
  4. Patients must have an established pediatrician within 90 miles of Stanford University for 3 years.
* Healthy Controls

  1. Age 4-18
  2. No psychiatric diagnosis

Exclusion Criteria:

* Any neuropsychiatric illness that may obscure the clear diagnosis of PANS

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The investigators to enroll 500 children with PANS/PANDAS and 100 healthy controls. Children's parents will also be enrolled to report information about their children as well as their own caregiver burden. The 500 patients with PANS will meet diagnostic criteria. These patients are targeted because this study is seeking to specifically assess the immunologic and neurological markers of PANS.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-03; Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Cerebral blood flow | Through study completion, up to 12 years
  The investigators will report results of altered cerebral blood flow from patients with PANS.
EEG patterns | Through study completion, up to 12 years
  The investigators will report results of abnormal EEG patterns from patients with PANS. All data will be obtained through the review of medical records, which are created during the routine clinical care of patients.
Rapid Eye Movement (REM) motor disinhibition | Through study completion, up to 12 years
  The investigators will report results of REM motor disinhibition from polysomnography studies. All data will be obtained through the review of medical records, which are created during the routine clinical care of patients.

SECONDARY OUTCOMES:
Global Impairment Scores | Every 2-4 weeks for up to 12 years
  All data will be obtained through the review of medical records, which are created during the routine clinical care of patients.
Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) | Every 2-4 weeks for up to 12 years
  All data will be obtained through the review of medical records, which are created during the routine clinical care of patients.
Columbia Impairment Scale | Every 2-4 weeks for up to 12 years
  All data will be obtained through the review of medical records, which are created during the routine clinical care of patients.
Caregiver Burden Inventory | Every 2-4 weeks for up to 12 years
  All data will be obtained through the review of medical records, which are created during the routine clinical care of patients.
Neurological findings | Every 2-4 weeks for up to 12 years
  The investigators will report data from neurological exam findings, including milk maid grip, chorea, choreiform movements of arms and legs, apraxia, overflow dystonia, truncal instability, piano-playing fingers, glabellar sign, etc. All data will be obtained through the review of medical records, which are created during the routine clinical care of patients. These results will be aggregated to report the number of participants with abnormal neurological findings.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data is available upon request as allowed by the Stanford Institutional Review board.

REFERENCES:
- [Background] Swedo SE, Leckman JF, Rose NR (2012) From Research Subgroup to Clinical Syndrome: Modifying the PANDAS Criteria to Describe PANS (Pediatric Acute-onset Neuropsychiatric Syndrome). Pediatr Therapeut 2:113. doi: 10.4172/2161-0665.1000113
- [Background] Chang K, Frankovich J, Cooperstock M, Cunningham MW, Latimer ME, Murphy TK, Pasternack M, Thienemann M, Williams K, Walter J, Swedo SE; PANS Collaborative Consortium. Clinical evaluation of youth with pediatric acute-onset neuropsychiatric syndrome (PANS): recommendations from the 2013 PANS Consensus Conference. J Child Adolesc Psychopharmacol. 2015 Feb;25(1):3-13. doi: 10.1089/cap.2014.0084. Epub 2014 Oct 17. PMID 25325534
- [Background] Murphy TK, Gerardi DM, Leckman JF. Pediatric acute-onset neuropsychiatric syndrome. Psychiatr Clin North Am. 2014 Sep;37(3):353-74. doi: 10.1016/j.psc.2014.06.001. PMID 25150567